CLINICAL TRIAL: NCT06980012
Title: Evaluation of the Impact of the Clinical Pharmacist in the Initiation and Follow-up of Oral Therapies in Oncology.
Brief Title: Evaluation of the Impact of the Clinical Pharmacist in Oral Therapies in Oncology.
Acronym: Pharmaimpact
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Polyclinique Lyon Nord (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-18-PLN
Record Dates: First submitted 2025-05-09; First posted 2025-05-20 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- specialized pharmaceutical consultation and follow-up in hospitals and community pharmacies (Experimental)
  Interventions: Procedure: Pharmaceutical consultation and follow-up
- specialized pharmaceutical consultation (Active Comparator)
  Interventions: Procedure: Pharmaceutical consultation

INTERVENTIONS:
Procedure: Pharmaceutical consultation — The pharmaceutical interview is a structured way of carrying out an optimized medication review with the patient. This interview takes place at the time of the first prescription of oral anti-cancer treatment.
  Arms: specialized pharmaceutical consultation
Procedure: Pharmaceutical consultation and follow-up — After the first prescription and at the treatment renewal date (+/- 2 days), the hospital pharmacist will contact the dispensing pharmacist to inform him/her of the patient's treatment, and then as part of the follow-up to detect any problems with treatment compliance (non-renewal of treatment by the patient, lack of follow-up, complaints of adverse effects by the patient). These events will be recorded in the observation book.
  Arms: specialized pharmaceutical consultation and follow-up in hospitals and community pharmacies

SUMMARY:
The hospital pharmacist plays a vital role at the time of the patient's first prescription in a healthcare facility, to inform the patient about his or her new therapy and create a link between the hospital and the patient's home pharmacy, so that the patient can continue to receive care at home. It is also essential that the hospital pharmacy and the patient's local pharmacy work together within a reasonable timeframe. This will help improve patient care and treatment follow-up, detect any undesirable effects and optimize their management..

The aim of this prospective interventional study is to measure the benefits of pharmaceutical monitoring in healthcare institutions at the initiation of oral therapy on patient compliance, side-effect management and adherence, in comparison with patients without this monitoring.

The primary endpoint is compliance with the Girerd questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from an oncological pathology (excluding hematological malignancies)
* Initiation of a specific treatment in the context of an oncological pathology: oral therapy treatment taken at home in oncology (which may follow surgery, radiotherapy or other in-patient treatments).
* Patient who has not yet started treatment or who has started treatment less than 30 days
* Patient with continuation of oral therapy dispensed in pharmacies

Exclusion Criteria:

* Patients suffering from hematological malignancies
* Patient living in an institution or hospital
* Patient under treatment for more than 30 days
* Patient undergoing treatment other than oral therapy (venous or subcutaneous anticancer treatment)
* Patient whose treatment after initiation is not dispensed in a pharmacy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Observance | 3 months and 6 months after treatment initiation
  The measurement of the primary endpoint is based on the use of a validated scale for assessing medication compliance: the Girerd scale. This is a 6-question questionnaire with a binary yes/no response. The score ranges from 0 to 6, with a "yes" worth 1 point.

CONTACTS AND LOCATIONS:
Locations (1):
- Polyclinique Lyon Nord, Rillieux-la-Pape, France

IPD SHARING:
Plan to Share IPD: No